CLINICAL TRIAL: NCT05700162
Title: The Effect of Showing Photographs, Videos and Live Images of Their Babies to Mothers During Milking on Breastmilk Amount, Mother-Infant Attachment and Breastfeeding Self-Efficacy Level: Randomized Controlled Experimental Study
Brief Title: The Effect of Showing Photographs, Videos and Live Images of Their Babies to Mothers During Milking
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Özlem MUMCU, Clinical Nurse Specialist, Eskisehir Osmangazi University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: EOU.SBE.OM.01
Record Dates: First submitted 2023-01-04; First posted 2023-01-26 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Breast Milk Expression; Breast Milk Collection; Mother-Infant Interaction
Keywords: prematüre; neonatal intensive care; breast milk
MeSH Terms: conditions — Breast Milk Expression | interventions — Moire Topography; Videotape Recording; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Photograph (Experimental): As soon as the mother starts to express her milk, she will be asked to look at the photo of her baby sent to her on whatsapp for 5 minutes.
  Interventions: Behavioral: Photograph
- Video (Experimental): As soon as the mother starts to express her milk, she will be asked to watch the 5-minute video of her baby sent to her on whatsapp.
  Interventions: Behavioral: Video
- Live Broadcast (Experimental): As soon as the mother starts to express her milk, she will be asked to watch the 5-minute live video of her baby with the call sent to her from WhatsApp.
  Interventions: Behavioral: Live Broadcast
- Control Group (Experimental): The mother will be asked to express both breasts for 15 minutes every 3 hours. No additional application will be made.
  Interventions: Behavioral: Control Group

INTERVENTIONS:
Behavioral: Photograph — As soon as she starts to express her milk from the mother, on whatsapp will be asked to look at the photo of the baby sent to her for 5 minutes. She will be asked to express both breasts for 15 minutes every 3 hours.
  Arms: Photograph
Behavioral: Video — As soon as the mother starts to express her milk, she will be asked to watch the 5-minute video of her baby sent to her on WhatsApp. She will be asked to express both breasts for 15 minutes every 3 hours.
  Arms: Video
Behavioral: Live Broadcast — As soon as the mother starts to express her milk, she will be asked to watch the 5-minute live video of her baby with the call sent to her from WhatsApp. She will be asked to express both breasts for 15 minutes every 3 hours.
  Arms: Live Broadcast
Behavioral: Control Group — She will be asked to express both breasts for 15 minutes every 3 hours. No additional action will be taken.
  Arms: Control Group

SUMMARY:
The study was planned to determine the effect of showing photographs, videos and live images of premature babies who could not be breastfed in the neonatal intensive care unit to their mothers on the amount of breast milk, mother-infant attachment and breastfeeding self-efficacy.

It is a randomized controlled experimental study.

DETAILED DESCRIPTION:
Separation of the baby from the mother, being admitted to the neonatal intensive care unit can quickly increase the mother's fears about her baby's health and appearance, it can be interpreted as a crisis for the family. When the baby is in the intensive care unit, it also becomes difficult for parents to participate in the care of the baby.

In this case, one of the negative emotions that parents often experience is anxiety.

In general, mothers experience more intense stress than fathers.The mother, who is away from her baby's care, feels tense, irritable and confused. She makes an effort to reach her baby, and when she fails to do so, she finds herself helpless and powerless. The neonatal intensive care nurse and the Women's Health nurse play a major role in the initiation of breastfeeding and the continuation of breastfeeding in pre-term newborns.

Early milking of mothers after premature birth increases breast milk production.

Despite early and frequent milking, some mothers may experience lower milk volume and milk production in the first few weeks. Therefore, mothers with premature babies should practice frequent breastfeeding/milking, massage and compression, hot application, acupuncture, yoga and relaxation exercises, etc., in order to increase prolactin secretion and increase breast milk production. focused on non-pharmacological methods such as. Another method that is considered effective is to show the mother a photo or video of the baby during milking. However, in the literature review, the number of available studies on this subject is only 2.

One of these studies was done in 2020. The other study was done in 2021. More work is needed on this subject. The aim of this study was to determine the effects of watching photos, videos and live images of babies during milking on the amount of breast milk, mother-infant attachment and breastfeeding self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Staying of the baby in the Neonatal Intensive Care Unit
* 34 weeks of gestation and below
* Mother's acceptance of the application
* The mother's inability to breastfeed her baby
* The mother has a smart mobile phone
* Mother's ability to read and write
* Being able to communicate with the mother (being able to read and write, speak Turkish, etc.)

Exclusion Criteria:

* Gestation week over 34
* The mother is breastfeeding her baby
* Being a smoker
* Having a systemic disease and constantly taking medication(s)
* Having a health problem that may affect the mother's milking (crack, mastitis, collapse etc.)

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2022-06-06 (Actual); Primary Completion 2024-08-08 (Estimated); Study Completion 2024-08-08 (Estimated)

PRIMARY OUTCOMES:
Mother-to-Infant Bonding Scale | up to 2 days
  It is a measurement tool that can be applied from the first day after birth and allows the mother to express her feelings towards her baby with a single word.
The Breastfeeding Self-Efficacy Scale: Psychometric Assessment of the Short Form | up to 2 days
  It consists of 33 items. It is a five-point Likert scale.

SECONDARY OUTCOMES:
Development of the breast milk expression experience measure | up to 2 days
  It consists of 11 items. It is a five-point Likert scale.

OTHER OUTCOMES:
Beck Anxiety Scale | 1 day
  It was developed by Beck et al. in 1988. It was aimed to measure the frequency of anxiety symptoms experienced.
Sleeplessness Severity Index | 1 day
  There are 7 questions in total. It is a tool for measuring the degree of insomnia.

CONTACTS AND LOCATIONS:
Overall Officials: Ayfer Açıkgöz, Study Director — ayferacikgoz u.edu.tr
Locations (1):
- Eskisehir Osmangazi Üniversity, Eskişehir, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No